CLINICAL TRIAL: NCT00128973
Title: Screening and Baseline Assessment of Patients With Abnormalities of Immune Function
Brief Title: Evaluation of Patients With Immune Function Abnormalities
Status: Recruiting | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 050213; 05-I-0213
Record Dates: First submitted 2005-08-09; First posted 2005-08-10 (Estimated); Last update posted 2026-01-05 (Actual); Status verified 2025-11-07

CONDITIONS: Chronic Granulomatous Disease (CGD); X-Linked Severe Combined Immune Deficiency (XSCID); Leukocyte Adhesion Deficiency 1 (LAD); Graft Versus Host Disease (cGvHD)
Keywords: Infection; Genetic; Inherited Disease; Immunity; Chronic; Abnormal Immune Function; Recurrent Infection; Chronic Granulomatous Disease; CGD; X-Linked Severe Combined Immune Deficiency (XSCID); XSCID; Leukocyte Adhesion Deficiency 1; LAD; Healthy Volunteer; HV
MeSH Terms: conditions — Granulomatous Disease, Chronic; Graft vs Host Disease; Bronchiolitis Obliterans Syndrome; Infections; Genetic Diseases, Inborn; Reinfection; X-Linked Combined Immunodeficiency Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy Volunteers: Healthy adult M/F 18-85 y/o.Hgb>=11.Wt>110 lbs. No heart,lung,kidney,bleeding disorders. No hep BorC since age 11. No IV drug use. No exposure to the AIDS virus. Not pregnant.
- Patients: Patients with abnormalities of immune function
- Relatives of Patient:: Relatives may be mother, father, siblings, children, grandparents, aunts, uncles, and first cousins to a patient.

SUMMARY:
This study will evaluate patients with abnormal immune function that results in recurrent or unusual infections or chronic inflammation. This may include inherited conditions, such as X-linked severe combined immunodeficiency (XSCID), chronic granulomatous disease (CGD), and leukocyte adhesion deficiency (LAD), or conditions resulting from outside factors, such as graft-versus-host disease (GVHD). The information from this study will be used to establish the pattern and pace of change of the disease and to help develop new treatments. The period of observation and study following enrollment in this study may be for up to one year. In addition these studies may provide the medical information needed to determine eligibility for enrollment in other clinical study protocols and more prolonged follow up.

Patients of any age with abnormal immune function who have recurrent or unusual infections, whose blood tests show evidence of immune dysfunction, or who have GVHD, XSCID, CGD or LAD may be eligible for this study. Patients' parents, siblings, grandparents, children, aunts, uncles and first cousins of any age also may be included. Healthy normal volunteers between 18 and 85 years of age are recruited as controls.

Normal volunteers undergo a physical examination and provide blood, saliva, and urine samples for immune function studies. Patients' family members provide a medical history, have a physical examination, and give blood and urine samples, and possibly a saliva sample. The samples are used for genetic and routine laboratory studies. Investigators may request tissue samples, such as biopsy specimens, previously removed for medical reasons to be sent to NIH for study. Patients undergo the following tests and procedures:

1. Medical history and physical examination.
2. Blood and urine tests, including analysis for genes involved in immune disorders.
3. Buccal smear (in some patients) for genetic studies. This involves scraping the lining of the mouth near the cheek.
4. Specialized tests to evaluate specific conditions in patients who have an immune disorder that might affect lung function, gum infections or eye problems. These may include chest x-ray, CT scan, breathing function test, dental, eye, and hearing examinations.
5. Follow-up visits of patients with immune problems may occur at 6 months and at one year after the first visit (or more frequently if medically required) to include:

   * Medical history update
   * Physical examination
   * Follow-up on abnormal test results and medical treatments initiated at NIH
   * Collection of blood, saliva, urine, or wound drainage samples for repeat immune function studies
   * Tissue study of specimens removed for medical reasons at other institutions besides NIH

DETAILED DESCRIPTION:
This protocol is designed for the screening and baseline assessment of and collection of research samples from patients with abnormalities of immune function as manifested by recurrent or unusual infections, recurrent or chronic inflammation, or previous laboratory evidence of immune dysfunction. After baseline assessments are complete, participants will remain on study to allow long-term assessments of the natural course of their condition. Abnormalities of immune function may be inherited or may be iatrogenic such as that following hematopoietic stem cell transplantation or other treatments resulting in prolonged immune dysfunction. Blood and/or bone marrow cells may also be used to investigate the utility of induced pluripotent stem cells (iPS) for immune cell derivation and targeted gene correction. This is not a protocol to study or screen for human immunodeficiency virus (HIV) infection, though patients with HIV infection who may have other causes for immune dysfunction are not excluded. First- or second-degree genetically related family members (limited to mother, father, siblings, grandparents, children, aunts, uncles, and first cousins of an affected patient) may also be screened for clinical, in vitro, and genetic correlates of immune abnormalities. Healthy Volunteers will be enrolled as a source of control blood samples for research testing, not to include genetic testing. Patients with documented immune dysfunction may receive limited medically indicated treatment if that medically indicated treatment is related to the abnormality of immune function under study. Results of clinically indicated diagnostic evaluations and treatments performed outside of this protocol may be collected for research use as part of this study. When screening and assessment is complete, patients will be offered an opportunity to participate in another study, or if there are no active studies appropriate for the patient, other options will be suggested to the primary or referring physician. Regardless of whether the patient enrolls on another NIH study, they will remain on this study for long-term follow-up of their condition.

This protocol will allow detailed long-term investigation of patients with abnormalities of immune function with the following goals:

1. To determine the degree, scope, and cause of immune dysfunction;
2. To establish the pace and pattern of change in the disease process;
3. To determine the extent of organ involvement and damage from immune dysfunction.

The assessments performed under this protocol are necessary to discover new causes of immune abnormalities, to delineate epidemiology of immune deficiencies, to develop new diagnostic and therapeutic tools, and to determine a patient s eligibility for other studies.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients:

To be eligible to participate in this study as a patient, an individual must meet the following criteria:

* Must be 2 years of age to be seen at the Clinical Center as an outpatient and they must not have any active infections. Send-in samples for clinical diagnosis at any age.
* Have an abnormality of immune function as manifested by:

  * recurrent or unusual infections,
  * recurrent or chronic inflammation, or
  * previous laboratory evidence of immune dysfunction.
* Have a primary physician outside of the NIH.

Relatives of Patient:

To be eligible to participate in this study as a patient relative, an individual must meet the following criteria:

* Be a biological mother, father, sibling, child, grandparent, aunt, uncle, or first cousin to a patient.

  --Sibling, child, first cousin, aunt, and uncle must be 2 years of age to be seen at the Clinical Center as an outpatient with no active infections, Send-in samples for clinical diagnosis at any age.
* Be willing to have blood stored for future studies and/or other research purposes.

Healthy Volunteers:

To be eligible to participate in this study as a healthy volunteer, an individual must meet the following criteria:

* Be a healthy adult of either sex and between age of 18 and 85 years old.
* Have a hemoglobin count of >=11.
* Weight greater than 110 pounds.
* Not have a history of intravenous injection drug use.
* Not have a history of engaging in high-risk activities for exposure to HIV.
* Be willing to have their blood samples stored for future research and modified to iPS cells.

EXCLUSION CRITERIA:

Patients and Relatives of Patient:

In general, there are no strict exclusion criteria for these cohorts. However, the presence of certain types of acquired abnormalities of immunity solely due to HIV, chemotherapeutic agent(s), or an underlying malignancy could be grounds for possible exclusion for a patient or relative of a patient. In the opinion of the investigator, the presence of such disease processes may interfere with evaluation of a co-existing abnormality of immunity that is the subject of study under this protocol. Pregnant females will not be allowed to participate in any procedure that may be dangerous to the pregnancy or the fetus.

Healthy Volunteers:

An individual who meets any of the following criteria will be excluded from participation as a healthy volunteer in this study:

* Have HIV or viral hepatitis (B or C), or history of viral hepatitis B or C since age 11.
* Receiving chemotherapeutic agent(s) or have underlying malignancy.
* Pregnant.
* Have history of heart, lung, kidney disease, or bleeding disorders.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Self referred, Physician referred
Sampling Method: Non-Probability Sample
Enrollment: 3500 (Estimated)
Dates: Start 2005-09-19 (Actual)

PRIMARY OUTCOMES:
To establish the pattern and pace of change of disease (frequency, distribution, type and extent of infections, inflammatory lesions and abnormalities of immune function) during a period of up to one year baseline assessment. | ongoing throughout study
  Identification pregression and pattern of disease over time
To establish the extent of organ involvement (infection and/or inflammation) and organ damage or dysfunction resulting from the abnormality of immune function. | ongoing throughout study
  Identification of severity of disease as it relates to immune function in PID
To determine genetic linkage and biochemical correlates of the patient s abnormality of immunity by study of first and second-degree related family members blood cells (buccal smears instead of blood for genetic studies in some individuals)... | ongoing throughout study
  Identification of genetic links and biochemical correlates of PID to clinical manifestations
To characterize the physiologic, biochemical or genetic basis of the abnormality of immunity. | ongoing throughout study
  Identification of the pathophysiology and genetic basis of abnormalities of immune function under study

SECONDARY OUTCOMES:
To establish a baseline assessment of the pace and extent of the disease before entering a therapeutic clinical trial. | ongoing throughout study
  Identification of best time with respect to disease process to place pts on a treatment protocol
To determine a patient s eligibility for other studies. | ongoing throughout study
  Patient recruitment to treatment protocols
To assess the patient s ability to safely tolerate specific aspects of other diagnostic or therapeutic research protocols. | ongoing throughout study
  Patients tolerate treatment for PID disease

CONTACTS AND LOCATIONS:
Overall Officials: Harry L Malech, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Noguchi M, Yi H, Rosenblatt HM, Filipovich AH, Adelstein S, Modi WS, McBride OW, Leonard WJ. Interleukin-2 receptor gamma chain mutation results in X-linked severe combined immunodeficiency in humans. Cell. 1993 Apr 9;73(1):147-57. doi: 10.1016/0092-8674(93)90167-o. PMID 8462096
- [Background] Puck JM, Deschenes SM, Porter JC, Dutra AS, Brown CJ, Willard HF, Henthorn PS. The interleukin-2 receptor gamma chain maps to Xq13.1 and is mutated in X-linked severe combined immunodeficiency, SCIDX1. Hum Mol Genet. 1993 Aug;2(8):1099-104. doi: 10.1093/hmg/2.8.1099. PMID 8401490
- [Background] Stephan JL, Vlekova V, Le Deist F, Blanche S, Donadieu J, De Saint-Basile G, Durandy A, Griscelli C, Fischer A. Severe combined immunodeficiency: a retrospective single-center study of clinical presentation and outcome in 117 patients. J Pediatr. 1993 Oct;123(4):564-72. doi: 10.1016/s0022-3476(05)80951-5. PMID 8410508
- [Derived] Strong J, Adhanom R, Kim CS, Saito Y, Meltzer JC, Hallaert P, Martinez S, Salancy A, Kong HH, Cowen EW, Castelo-Soccio L, Murphy PM, McDermott DH, Brownell I. Risk of Superficial Fungal Infections in WHIM Syndrome. Dermatol Ther (Heidelb). 2025 May;15(5):1173-1179. doi: 10.1007/s13555-025-01396-0. Epub 2025 Apr 3. PMID 40178760
- [Derived] De Ravin SS, Cowen EW, Zarember KA, Whiting-Theobald NL, Kuhns DB, Sandler NG, Douek DC, Pittaluga S, Poliani PL, Lee YN, Notarangelo LD, Wang L, Alt FW, Kang EM, Milner JD, Niemela JE, Fontana-Penn M, Sinal SH, Malech HL. Hypomorphic Rag mutations can cause destructive midline granulomatous disease. Blood. 2010 Aug 26;116(8):1263-71. doi: 10.1182/blood-2010-02-267583. Epub 2010 May 20. PMID 20489056
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2005-I-0213.html